CLINICAL TRIAL: NCT04098393
Title: A Pilot Study of Condensed Busulfan, Melphalan, and Fludarabine Conditioning Prior to Ex-vivo CD34+ Selected Allogeneic Hematopoietic Cell Transplantation
Brief Title: Giving Chemotherapy for a Shortened Amount of Time Before a Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-245
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Hematologic Malignancies
Keywords: Busulfan; Melphalan; Fludarabine; Allogeneic Hematopoietic Cell Transplantation; 19-245
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Busulfan; fludarabine; Melphalan; Antilymphocyte Serum

STUDY DESIGN:
Intervention Model Description: This is a pilot study in which adult patients with hematologic malignancies undergoing ex-vivo CD34-selected allo-HCT will receive a condensed version of our standard bu/mel/flu regimen, reducing the length of the conditioning regimen from 8 days to 5 days.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- patients hematologic malignancies other than multiple myeloma (Experimental): A. Busulfan 3.2 mg/kg/day, with dose adjustments made according to pharmacokinetic (PK) levels. B. Melphalan (70mg/m2/day) administered on days -6 and -5. C. Fludarabine (25mg/m2/ day) administered on days -6, -5, -4, -3, and -2. All patients receiving matched related or unrelated donor allografts receive anti-thymocyte globulin (ATG) 2.5 mg/kg/day on days -3 and -2 to deplete chemotherapy resistant host T-cells that could hinder engraftment, and it may provide additional GVHD prophylaxis.
  Interventions: Drug: Busulfan 3.2 mg/kg/day; Drug: Fludarabine; Drug: Melphalan; Drug: Antithymocyte globulin (ATG); Procedure: Allogeneic hematopoietic cell transplantation (Allo-HCT)
- patients with multiple myeloma (Experimental): A. Busulfan 0.8 mg/kg every 6 hours x 10 doses, with dose adjustments made according to PK levels. B. Melphalan (70 mg/m2/day) administered on days -6 and -5. C. Fludarabine (25 mg/m2/day) administered on days -6, -5, -4, -3, -2. All patients receiving matched related or unrelated donor allografts receive anti-thymocyte globulin (ATG) 2.5 mg/kg/day on days -3 and -2 to deplete chemotherapy resistant host T-cells that could hinder engraftment, and it may provide additional GVHD prophylaxis.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Antithymocyte globulin (ATG); Drug: Busulfan 0.8 mg/kg; Procedure: Allogeneic hematopoietic cell transplantation (Allo-HCT)

INTERVENTIONS:
Drug: Busulfan 3.2 mg/kg/day — Busulfan 3.2 mg/kg/day, with dose adjustments made according to pharmacokinetic (PK) levels.
  Arms: patients hematologic malignancies other than multiple myeloma
Drug: Fludarabine — Fludarabine (25mg/m2/ day) administered on days -6, -5, -4, -3, and -2.
Drug: Melphalan — Melphalan (70mg/m2/day) administered on days -6 and -5.
Drug: Antithymocyte globulin (ATG) — ATG will be given based on a dynamic nomogram based on the patient's absolute lymphocyte count at the start of conditioning and can result in 2 or 3 days of ATG administration.
Drug: Busulfan 0.8 mg/kg — Busulfan 0.8 mg/kg every 6 hours x 10 doses, with dose adjustments made according to PK levels.
  Arms: patients with multiple myeloma
Procedure: Allogeneic hematopoietic cell transplantation (Allo-HCT) — Allogeneic hematopoietic cell transplantation following the conditioning regimen.

SUMMARY:
The purpose of this study is to see if a condensed version of the chemotherapy regimen busulfan, melphalan, fludarabine (bu/mel/flu) and the drug antithymocyte globulin (ATG-also referred to as rATG or thymoglobulin) can have the same or fewer number of severe side effects in people with various blood cancers 30 days after they receive an allogeneic hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old.
* Patients with any of the following hematologic malignancies for which allo-HCT is indicated, including:

  * Acute myeloid leukemia (AML) with intermediate or high-risk features in CR1.
  * Relapsed AML in ≥ CR2.
  * Acute leukemias of ambiguous lineage in ≥ CR1.
  * Acute lymphoid leukemia (ALL) in CR1 with clinical, flow cytometric, or molecular features indicating a high risk for relapse, or ALL in ≥ CR2.
  * CML meeting one of the following criteria:
  * Failed response to or intolerant to BCR-ABL tyrosine kinase inhibitors (TKIs).
  * CML with BCR-ABL mutation consistent with poor response to TKIs (e.g., T315I mutation)
  * CML in accelerated phase or blast crisis with <10% blasts after therapy, or in second chronic phase.
  * Myelodysplastic syndromes (MDS), myeloproliferative neoplasms (MPN), or MDS/MPN overlap syndromes with least one of the following:
  * Revised International Prognostic Scoring System risk score of intermediate or higher at the time of transplant evaluation.
  * Life-threatening cytopenias.
  * Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype.
  * Therapy related disease or disease evolving from other malignant processes.
  * Chronic myelomonocytic leukemia (CMML-1 or CMML-2).
  * Severe aplastic anemia.
  * Relapsed Hodgkin lymphoma meeting both of the following criteria:
  * Responding to therapy prior to enrollment.
  * Relapse after autologous HCT or are ineligible for autologous HCT.
  * Relapsed non-Hodgkin lymphoma meeting both of the following criteria:
  * Responding to therapy prior to enrollment.
  * Relapse after prior autologous HCT or are ineligible for autologous HCT.
  * High-risk multiple myeloma following autologous HCT or relapsed multiple myeloma following autologous HCT with chemosensitive disease.
* Adequate organ function is required, defined as follows:

  * Serum bilirubin ≤ 2 mg/dL, unless benign congenital hyperbilirubinemia. Patients with hyperbilirubinemia related to paroxysmal nocturnal hemoglobinuria or other hemolytic disorders are eligible with PI approval.
  * AST, ALT, and alkaline phosphatase < 3 times the upper limit of normal unless thought to be disease-related.
  * Creatinine clearance ≥ 50 ml/min (calculated by Cockcroft Gault)
  * LVEF ≥ 45% by MUGA or resting echocardiogram.
  * Pulmonary function (FEV1 and corrected DLCO) ≥ 50% predicted.
* Adequate performance status of ECOG ≤ 2.
* Each patient must be willing to participate as a research subject and must sign an informed consent form.

Exclusion Criteria:

* Patients with active extramedullary disease.
* Patients with active central nervous system malignancy.
* Active and/or uncontrolled infection at the time of allo-HCT.
* Patients who have undergone previous allo-HCT.
* Patients who have undergone previous autologous HCT within the last 6 months, with the exclusion of high-risk multiple myeloma patients.
* Patient seropositivity for HIV I/II and/or HTLV I/II.
* Females who are pregnant or breastfeeding.
* Patients unwilling to use contraception during the study period.
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol.

Donor Inclusion and Exclusion Criteria:

* Must be a 10/10 HLA genotypically matched related or unrelated donor at A, B, C, DRB1, and DQB1 loci, as tested by DNA analysis.
* Able to provide informed consent for the donation process per institutional standards.
* Meet standard criteria for donor collection as defined by the National Marrow Donor Program Guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
the number of grade 4 toxicities | in the first 30 days post-HCT
  All grade 4 CTCAEv5.0 toxicities are included except for hematologic toxicities that are considered expected for patients receiving myeloablative conditioning.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scordo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm